CLINICAL TRIAL: NCT06682559
Title: Comparison of Two Different Healing Abutments in Single Posterior Implants: A Randomized Clinical Trial
Brief Title: Comparison Between Two Different Healing Abutments in Single Posterior Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rania Elsayed, Principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0991-10
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Dental Implants; Dental Implants, Single-tooth
Keywords: Dental implants; single missing posterior teeth; peri-implant soft tissues

STUDY DESIGN:
Who Masked: Participant
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prefabricated healing abutment with scan peg (Neoss implant system, Harrogate, England) (Experimental): 12 participants will receive single posterior implants by fully guided implant protocol followed by placement of prefabricated healing abutment with scan peg having convex emergence profile
  Interventions: Other: Prefabricated healing abutment with scan peg
- Customized healing abutment (Active Comparator): 12 participants will receive single posterior implants by fully guided implant protocol followed by placement of custom healing abutment having concave emergence profile
  Interventions: Other: Customized healing abutment

INTERVENTIONS:
Other: Prefabricated healing abutment with scan peg — 12 participants will receive single posterior implants by fully guided implant protocol followed by placement of prefabricated healing abutment with scan peg having convex emergence profile
  Arms: Prefabricated healing abutment with scan peg (Neoss implant system, Harrogate, England)
Other: Customized healing abutment — 12 participants will receive single posterior implants by fully guided implant protocol followed by placement of custom healing abutment having concave emergence profile
  Arms: Customized healing abutment

SUMMARY:
The aim of this randomized clinical trial is to evaluate the volumetric analysis of peri-implant soft tissues after 3 months of the use of a prefabricated healing abutment with scan peg in comparison to customized healing abutment.

DETAILED DESCRIPTION:
Volumetric analysis of peri-implant soft tissues after 3 months of the use of a prefabricated healing abutment with scan peg with convex emergence profile in comparison to customized healing abutment with concave emergence profile.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are classified as ASA I or II physical status and require mandibular single implants (single missing mandibular posterior teeth) with:

  1. Proper bone height and width.
  2. Adequate zone of keratinized tissue (at least 2 mm)

Exclusion Criteria:

* Any systematic disease as uncontrolled diabetes mellitus or metabolic bone diseases
* Pregnancy and Lactation
* A history of head and neck radiation treatment.
* Chronic periodontal diseases.
* Poor oral hygiene (Silness-Löe plaque index score 2 and 3)
* Parafunctional habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of peri-implant soft tissues volume | 3 months
  Each participant will undergo volumetric analysis of peri-implant soft tissues after 3 months healing either after using prefabricated healing abutment with scan peg in comparison to customized healing abutment using a 3D meteorology software (GOM inspect). It will be measured in millimeter cube

CONTACTS AND LOCATIONS:
Overall Officials: Mervat E Abdellah, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided